CLINICAL TRIAL: NCT06501339
Title: Maintenance Electroconvulsive Therapy (ECT) Versus Aripiprazole on Psychopathology and Cerebral Perfusion in Clozapine-resistant Schizophrenia: a Randomized, Double-blind Controlled Trial
Brief Title: Maintenance Electroconvulsive Therapy (ECT) Versus Aripiprazole in Clozapine-resistant Schizophrenia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, BISWA RANJAN MISHRA, Additional Professor, Psychiatry, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T/EMF/Psych/23-24/13
Record Dates: First submitted 2023-10-14; First posted 2024-07-15 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Clozapine Resistant Schizophrenia
Keywords: Clozapine resistant; schizophrenia; Aripiprazole; m-ECT
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maintenance ECT (Experimental)
  Interventions: Procedure: maintenance ECT
- Aripiprazole (Active Comparator)
  Interventions: Drug: Aripiprazole tablet

INTERVENTIONS:
Procedure: maintenance ECT — Frequency of weekly sessions for 1 month, then fortnightly for 5 months
  Arms: Maintenance ECT
Drug: Aripiprazole tablet — Aripiprazole 10 mg in the morning throughout the study period
  Arms: Aripiprazole

SUMMARY:
The pharmacological treatment options in schizophrenia developing resistance to clozapine are limited. Few studies have found ECT as beneficial in TRS, including CRS. However, literature on the role of M-ECT in maintaining the therapeutic gains of acute ECT in CRS is lacking. The objective of the study is to compare the efficacy of M-ECT vs aripiprazole as an add-on to ongoing clozapine on the severity of symptom dimensions, cerebral perfusion, global functioning and cognitions in patients with CRS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients clinically diagnosed with CRS (currently under clozapine)
2. Patients aged 18-60 years of either sex.
3. LAR giving voluntary written consent for participation in the study

Exclusion Criteria:

1. Patient already on ECT or aripiprazole.
2. History of psychoactive substance abuse or dependence.
3. Co-morbid psychiatric, major medical or neurological disorders.
4. History of organicity or significant head injury.
5. Pacemaker or metal in any body part, excluding the mouth. Pregnant and breastfeeding females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Positive And Negative Syndome Scale score | Baseline, 6 weeks, 12 weeks, 24 weeks
  Change from baseline in Total, Positive, negative and general scores with treatment. Minimum value: 30; maximum value: 210. Higher score means worsening of symptoms

SECONDARY OUTCOMES:
Change in regional cerebral blood flow by the SPECT-CT brain | Baseline, 24 weeks
  Change frome baseline in regional cerebral blood flow by the SPECT-CT brain with treatment
change in the Monteal Cognitive Assessment scores | Baseline,6 weeks, 12 weeks, 24 weeks
  change from baseline in the Monteal Cognitive Assessment scores with treatment. Minimum Value: 0 Maximum Value: 30: Higher score indicate better cognitive function
change in the Global Assessment of Functioning scores | Baseline, 6 weeks, 12 weeks, 24 weeks
  change from baseline in the Global Assessment of Functioning scores with treatment Minimum Value: 0 Maximum Value: 100: Higher score indicate better global functioning
Safety evaluation | Baseline,6 weeks, 12 weeks, 24 weeks
  Number of events observed in each patient and patients with at least one adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Rituparna Maiti, MD, Study Director — AIIMS Bhubaneswar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siskind D, Orr S, Sinha S, Yu O, Brijball B, Warren N, MacCabe JH, Smart SE, Kisely S. Rates of treatment-resistant schizophrenia from first-episode cohorts: systematic review and meta-analysis. Br J Psychiatry. 2022 Mar;220(3):115-120. doi: 10.1192/bjp.2021.61. PMID 35049446
- [Background] Siskind D, Siskind V, Kisely S. Clozapine Response Rates among People with Treatment-Resistant Schizophrenia: Data from a Systematic Review and Meta-Analysis. Can J Psychiatry. 2017 Nov;62(11):772-777. doi: 10.1177/0706743717718167. Epub 2017 Jun 28. PMID 28655284
- [Background] Campana M, Falkai P, Siskind D, Hasan A, Wagner E. Characteristics and definitions of ultra-treatment-resistant schizophrenia - A systematic review and meta-analysis. Schizophr Res. 2021 Feb;228:218-226. doi: 10.1016/j.schres.2020.12.002. Epub 2021 Jan 14. PMID 33454644
- [Background] Rey JM, Walter G. Half a century of ECT use in young people. Am J Psychiatry. 1997 May;154(5):595-602. doi: 10.1176/ajp.154.5.595. PMID 9137112
- [Background] Chanpattana W, Andrade C. ECT for treatment-resistant schizophrenia: a response from the far East to the UK. NICE report. J ECT. 2006 Mar;22(1):4-12. doi: 10.1097/00124509-200603000-00002. PMID 16633199